CLINICAL TRIAL: NCT02773771
Title: Strategies to Reduce Organic Muscle Atrophy in the Intensive Care Unit (STROMA-ICU)
Brief Title: Strategies to Reduce Organic Muscle Atrophy in the Intensive Care Unit
Acronym: STROMA-ICU
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Per IRB submission history, submission declined and withdrawn. PI no longer at institution.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016p001044
Record Dates: First submitted 2016-05-05; First posted 2016-05-16 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Muscle Atrophy
Keywords: Muscle Atrophy; Critical Illness; Ultrasound; beta-hydroxy-beta-methylbutyrate; ICU
MeSH Terms: conditions — Muscular Atrophy; Critical Illness | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + Vital HP (Placebo Comparator): GROUP 1 will receive Placebo (within 24 hours of ICU admission) and Vital HP ® (while on tube feeds). Vital HP® is on the Massachusetts General hospital formulary, but it is often restricted to patients with malabsorption due to its higher cost compared to other standard enteral nutrition formulas.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vital HP®
- B-hydroxy-B-methylbutyrate (HMB) + Vital HP (Experimental): GROUP 2 will receive beta-hydroxy-beta-methylbutyrate (within 24 hours of ICU admission) and Vital HP ® (while on tube feeds). Vital HP® is on the Massachusetts General hospital formulary, but it is often restricted to patients with malabsorption due to its higher cost compared to other standard enteral nutrition formulas. The investigators will limit HMB dosing to 3g/day since this is the most widely studied dose.
  Interventions: Dietary Supplement: beta-hydroxy-beta-methylbutyrate; Dietary Supplement: Vital HP®

INTERVENTIONS:
Dietary Supplement: beta-hydroxy-beta-methylbutyrate — HMB is a leucine metabolite that may also be a potent mediator of anabolic processes in skeletal muscle; subjects will not receive >3g of HMB/ day.
  Other Names: HMB
  Arms: B-hydroxy-B-methylbutyrate (HMB) + Vital HP
Dietary Supplement: Placebo — The placebo is cornstarch and will be mixed in with Vital HP. The solution will look identical to the intervention arm.
  Arms: Placebo + Vital HP
Dietary Supplement: Vital HP® — Vital HP® is a form of enteral nutrition a part of the Massachusetts General enteral formulary

SUMMARY:
Acute muscle wasting occurs early and rapidly during the first week of critical illness and contributes substantially to weakness acquired in the ICU. Muscle wasting and subsequent weakness is associated with delayed liberation from mechanical ventilation, prolonged hospital length of stay, long-term functional disability, and worse quality of life. Moreover, low muscle volume as well as ICU-acquired weakness increases the risk of mortality in critically ill patients. Although several factors likely accelerate skeletal muscle wasting during critical illness (e.g., immobility, inflammation, multi-organ failure), the understanding of the underlying mechanisms remains limited and is reflected in the lack of effective interventions to prevent the loss of muscle mass in ICU patients. To-date, there is no known safe and effective pharmacological or nutritional intervention to attenuate the acute loss of muscle mass in ICU patients.

Leucine is an amino acid widely regarded for its anabolic effects on muscle metabolism. However, the concentrations required to maximize its anti-proteolytic effects are far greater than the concentrations required to maximally stimulate protein synthesis. This has resulted in the search for leucine metabolites that may also be potent mediators of anabolic processes in skeletal muscle; one such compound is β-hydroxy-β-methylbutyrate (HMB). HMB is thought to primarily facilitate protein synthesis through stimulation of mammalian target of rapamycin (mTOR), a protein kinase responsive to mechanical, hormonal, and nutritional stimuli that plays a central role in the control of cell growth. Randomized, controlled trials to assess the effect of HMB supplementation on clinical outcomes in patients with chronic diseases are limited, and even fewer studies have assessed its effects on skeletal muscle metabolism during critical illness. Furthermore, despite compelling preclinical evidence, the exact mechanisms underlying the effect of HMB supplementation during acute catabolic stress in humans is not well defined. Therefore, the investigators goal is to study the impact of early HMB supplementation on skeletal muscle mass in ICU patients and to explore the mechanisms by which HMB may exert its effects on skeletal muscle metabolism during critical illness.

DETAILED DESCRIPTION:
Acute muscle wasting occurs early and rapidly during the first week of critical illness and contributes substantially to weakness acquired in the ICU. Muscle wasting and subsequent weakness is associated with delayed liberation from mechanical ventilation, prolonged hospital length of stay (LOS), long-term functional disability, and worse quality of life. Moreover, low muscle volume and ICU-acquired weakness increases the risk of mortality in critically ill patients. Although several factors likely accelerate skeletal muscle wasting during critical illness (e.g., immobility, muscle unloading, inflammation, multi-organ failure), the understanding of the underlying mechanisms remains limited and is reflected in the lack of effective interventions to prevent the loss of muscle mass in ICU patients.

Muscle mass is maintained through balanced protein breakdown and synthesis . As such, for wasting to occur, catabolic pathways must be increased relative to anabolic processes. In general, nutritional status is an important factor for maintaining skeletal muscle homeostasis. However, adequate caloric delivery is often challenging in ICU patients and recent data suggest that high protein delivery in early critical illness may adversely impact muscle protein synthesis. Moreover, randomized, placebo-controlled, clinical trials (RCTs) in ICU patients do not support the use of aggressive early macronutrient delivery. Such findings emphasize the need for targeted therapies to enhance anabolic pathways, which may improve clinical outcomes in critically ill patients.

The amino acid leucine is widely regarded for its anabolic effects on muscle metabolism, but the concentrations required to maximize its anti-proteolytic effects are far greater than the concentrations required to maximally stimulate protein synthesis. This has resulted in the search for leucine metabolites that may also be potent mediators of anabolic processes in skeletal muscle -- one such compound is β-hydroxy-β-methylbutyrate (HMB).

HMB is thought to primarily facilitate protein synthesis through stimulation of mammalian target of rapamycin (mTOR), a protein kinase responsive to mechanical, hormonal, and nutritional stimuli that plays a central role in the control of cell growth. Indeed, preclinical studies demonstrate that HMB supplementation increases phosphorylation of mTOR as well as its downstream targets. Preclinical data also suggest that HMB supplementation results in an increase in skeletal muscle insulin-like growth factor 1(IGF-1) levels, which may further stimulate mTOR. In addition, HMB may influence systemic levels of myostatin, a key negative regulator of mature skeletal muscle growth. Myostatin has been shown to reduce muscle protein synthesis by inhibiting mTOR signaling and by increasing proteolytic mechanisms. Recent preclinical data suggest that HMB may reduce myostatin levels and attenuate skeletal muscle atrophy. Furthermore, preclinical data has shown that HMB also stimulates the release of irisin, a newly discovered myokine, which up-regulates IGF-1 and inhibits myostatin.

On the other hand, skeletal muscle proteolysis is thought to occur primarily through the ubiquitin-proteasome system, which is an energy-dependent proteolytic system that degrades intracellular proteins. The activity of this pathway is thought to be regulated through expression of nuclear factor kappa B (NF-κB), which is significantly increased in conditions such as fasting, immobilization, bed rest, and in various disease states. In preclinical studies, HMB has been shown to decrease proteasome expression and reduce activity of this pathway during catabolic states. Furthermore, caspase proteases (in particular, caspase protease-3 and caspase protease-9) are thought to induce skeletal muscle proteolysis through apoptosis of myonuclei. Preclinical data suggest that in catabolic states, HMB attenuates the up-regulation of caspases, which in turn, reduces myonuclear apoptosis and reduces skeletal muscle protein degradation.

Randomized controlled trials (RCTs) that have assessed the effect of HMB supplementation on clinical outcomes in patients with chronic diseases are limited, and even fewer studies have assessed its effects on skeletal muscle metabolism during critical illness. Furthermore, despite compelling preclinical evidence, the exact mechanisms underlying the effect of HMB supplementation during acute catabolic stress in humans is not well defined.

Therefore, the investigators goal is to study the impact of early HMB supplementation on skeletal muscle mass in surgical ICU patients and to explore the mechanisms by which HMB may exert beneficial effects on skeletal muscle metabolism during the course of critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. English-speaking
3. Expected to require at least 72 hours of ICU care
4. Able to provide written/verbal consent or have a suitable healthcare proxy
5. Able to ultrasound the diaphragm and quadriceps muscles in a consistent location for 7 days
6. Ability to take study drug orally vs. an indwelling nasogastric, orogastric, gastric, or gastrojejunostomy tube

Exclusion Criteria:

1. Pregnant or peri-partum female
2. Baseline hemoglobin less than 8g/dL
3. Not expected to survive beyond 72 hours
4. Unable to provide a written/verbal consent or an available healthcare proxy
5. Enrolled in another study which may interfere with the current study
6. Prior ICU admission with 1 year of current admission or more than 7 days of hospital admission before transfer to the ICU
7. Strict "nil per os" (NPO) status
8. High output through naso/orogastric tube
9. Clinically significant bowel obstruction
10. Active cancer (except for actinic keratosis, squamous cell carcinoma, and basal cell carcinoma confined to the skin)
11. Palliative care status
12. Known or anticipated history of difficult blood draws
13. History of elevated low density lipoprotein (LDL) and not on a stable treatment regimen
14. Blood urea nitrogen (BUN): creatinine >20 without an underlying cause
15. History of hypoglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in muscle thickness (diaphragm) at 14 days after ICU admission. | Day 14 of ICU admission or through study completion, an average of 1 month
  Change in muscle thickness will be assessed via ultrasound (base line and 14 days)
Change in muscle thickness (quadriceps at 14 days after ICU admission. | Day 14 of ICU admission or through study completion, an average of 1 month
  Change in muscle thickness will be assessed via ultrasound (baseline and 14 days)

SECONDARY OUTCOMES:
Intensive care unit length of stay | Time of admission to the ICU until the time of discharge from the intensive care unit, up to 100 weeks
Hospital Length of Stay | Time of discharge from the ICU until hospital discharge, up to 100 weeks
30-day ventilator free days | number of days during ICU admission not requiring invasive mechanical ventilation support, or until study completion, up to 100 weeks
  number of days not requiring invasive mechanical ventilation support
Discharge destination (home vs. non-home) | time of discharge until 90 days after discharge
  Assess where patients as discharged to
30-day readmission | From the time of hospital discharge until 30-days after hospitalization
  Assess readmission rates in both groups
30-day all-cause mortality | From the time of hospital discharge until 30 days after hospitalization
  Assess 30 day all cause mortality in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A. Quraishi, MD,MHA,MMSc, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Griffiths RD, Hall JB. Exploring intensive care unit-acquired weakness. Preface. Crit Care Med. 2009 Oct;37(10 Suppl):S295. doi: 10.1097/CCM.0b013e3181b6f411. No abstract available. PMID 20046112
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Stevens RD, Dowdy DW, Michaels RK, Mendez-Tellez PA, Pronovost PJ, Needham DM. Neuromuscular dysfunction acquired in critical illness: a systematic review. Intensive Care Med. 2007 Nov;33(11):1876-91. doi: 10.1007/s00134-007-0772-2. Epub 2007 Jul 17. PMID 17639340
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] Puthucheary ZA, Hart N. Skeletal muscle mass and mortality - but what about functional outcome? Crit Care. 2014 Feb 17;18(1):110. doi: 10.1186/cc13729. PMID 24528611
- [Background] Lee JJ, Waak K, Grosse-Sundrup M, Xue F, Lee J, Chipman D, Ryan C, Bittner EA, Schmidt U, Eikermann M. Global muscle strength but not grip strength predicts mortality and length of stay in a general population in a surgical intensive care unit. Phys Ther. 2012 Dec;92(12):1546-55. doi: 10.2522/ptj.20110403. Epub 2012 Sep 13. PMID 22976446
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Weijs PJ, Looijaard WG, Dekker IM, Stapel SN, Girbes AR, Oudemans-van Straaten HM, Beishuizen A. Low skeletal muscle area is a risk factor for mortality in mechanically ventilated critically ill patients. Crit Care. 2014 Jan 13;18(2):R12. doi: 10.1186/cc13189. PMID 24410863
- [Background] Plank LD, Hill GL. Similarity of changes in body composition in intensive care patients following severe sepsis or major blunt injury. Ann N Y Acad Sci. 2000 May;904:592-602. doi: 10.1111/j.1749-6632.2000.tb06521.x. PMID 10865810
- [Background] Puthucheary Z, Montgomery H, Moxham J, Harridge S, Hart N. Structure to function: muscle failure in critically ill patients. J Physiol. 2010 Dec 1;588(Pt 23):4641-8. doi: 10.1113/jphysiol.2010.197632. Epub 2010 Oct 20. PMID 20961998
- [Background] Vanhorebeek I, Van den Berghe G. Hormonal and metabolic strategies to attenuate catabolism in critically ill patients. Curr Opin Pharmacol. 2004 Dec;4(6):621-8. doi: 10.1016/j.coph.2004.07.007. PMID 15525554
- [Background] Thibault R, Pichard C. Nutrition and clinical outcome in intensive care patients. Curr Opin Clin Nutr Metab Care. 2010 Mar;13(2):177-83. doi: 10.1097/MCO.0b013e32833574b9. PMID 19996743
- [Background] Bear DE, Puthucheary ZA, Hart N. Early feeding during critical illness. Lancet Respir Med. 2014 Jan;2(1):15-7. doi: 10.1016/S2213-2600(13)70262-5. Epub 2013 Dec 23. No abstract available. PMID 24461888
- [Background] Peev MP, Yeh DD, Quraishi SA, Osler P, Chang Y, Gillis E, Albano CE, Darak S, Velmahos GC. Causes and consequences of interrupted enteral nutrition: a prospective observational study in critically ill surgical patients. JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):21-7. doi: 10.1177/0148607114526887. Epub 2014 Apr 7. PMID 24714361
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Hermans G, Casaer MP, Clerckx B, Guiza F, Vanhullebusch T, Derde S, Meersseman P, Derese I, Mesotten D, Wouters PJ, Van Cromphaut S, Debaveye Y, Gosselink R, Gunst J, Wilmer A, Van den Berghe G, Vanhorebeek I. Effect of tolerating macronutrient deficit on the development of intensive-care unit acquired weakness: a subanalysis of the EPaNIC trial. Lancet Respir Med. 2013 Oct;1(8):621-629. doi: 10.1016/S2213-2600(13)70183-8. Epub 2013 Sep 10. PMID 24461665
- [Background] Casaer MP, Wilmer A, Hermans G, Wouters PJ, Mesotten D, Van den Berghe G. Role of disease and macronutrient dose in the randomized controlled EPaNIC trial: a post hoc analysis. Am J Respir Crit Care Med. 2013 Feb 1;187(3):247-55. doi: 10.1164/rccm.201206-0999OC. Epub 2012 Nov 29. PMID 23204255
- [Background] Doig GS, Simpson F; Early PN Trial Investigators Group. Early parenteral nutrition in critically ill patients with short-term relative contraindications to early enteral nutrition: a full economic analysis of a multicenter randomized controlled trial based on US costs. Clinicoecon Outcomes Res. 2013 Jul 22;5:369-79. doi: 10.2147/CEOR.S48821. Print 2013. PMID 23901287
- [Background] Wilson JM, Fitschen PJ, Campbell B, Wilson GJ, Zanchi N, Taylor L, Wilborn C, Kalman DS, Stout JR, Hoffman JR, Ziegenfuss TN, Lopez HL, Kreider RB, Smith-Ryan AE, Antonio J. International Society of Sports Nutrition Position Stand: beta-hydroxy-beta-methylbutyrate (HMB). J Int Soc Sports Nutr. 2013 Feb 2;10(1):6. doi: 10.1186/1550-2783-10-6. PMID 23374455
- [Background] Zanchi NE, Nicastro H, Lancha AH Jr. Potential antiproteolytic effects of L-leucine: observations of in vitro and in vivo studies. Nutr Metab (Lond). 2008 Jul 17;5:20. doi: 10.1186/1743-7075-5-20. PMID 18637185
- [Background] Eley HL, Russell ST, Baxter JH, Mukerji P, Tisdale MJ. Signaling pathways initiated by beta-hydroxy-beta-methylbutyrate to attenuate the depression of protein synthesis in skeletal muscle in response to cachectic stimuli. Am J Physiol Endocrinol Metab. 2007 Oct;293(4):E923-31. doi: 10.1152/ajpendo.00314.2007. Epub 2007 Jul 3. PMID 17609254
- [Background] Aversa Z, Bonetto A, Costelli P, Minero VG, Penna F, Baccino FM, Lucia S, Rossi Fanelli F, Muscaritoli M. beta-hydroxy-beta-methylbutyrate (HMB) attenuates muscle and body weight loss in experimental cancer cachexia. Int J Oncol. 2011 Mar;38(3):713-20. doi: 10.3892/ijo.2010.885. Epub 2010 Dec 23. PMID 21184031
- [Background] Gerlinger-Romero F, Guimaraes-Ferreira L, Giannocco G, Nunes MT. Chronic supplementation of beta-hydroxy-beta methylbutyrate (HMbeta) increases the activity of the GH/IGF-I axis and induces hyperinsulinemia in rats. Growth Horm IGF Res. 2011 Apr;21(2):57-62. doi: 10.1016/j.ghir.2010.12.006. Epub 2011 Jan 14. PMID 21237681
- [Background] Kornasio R, Riederer I, Butler-Browne G, Mouly V, Uni Z, Halevy O. Beta-hydroxy-beta-methylbutyrate (HMB) stimulates myogenic cell proliferation, differentiation and survival via the MAPK/ERK and PI3K/Akt pathways. Biochim Biophys Acta. 2009 May;1793(5):755-63. doi: 10.1016/j.bbamcr.2008.12.017. Epub 2009 Jan 3. PMID 19211028
- [Background] Goodman CA, McNally RM, Hoffmann FM, Hornberger TA. Smad3 induces atrogin-1, inhibits mTOR and protein synthesis, and promotes muscle atrophy in vivo. Mol Endocrinol. 2013 Nov;27(11):1946-57. doi: 10.1210/me.2013-1194. Epub 2013 Sep 3. PMID 24002653
- [Background] Mobley CB, Fox CD, Ferguson BS, Amin RH, Dalbo VJ, Baier S, Rathmacher JA, Wilson JM, Roberts MD. L-leucine, beta-hydroxy-beta-methylbutyric acid (HMB) and creatine monohydrate prevent myostatin-induced Akirin-1/Mighty mRNA down-regulation and myotube atrophy. J Int Soc Sports Nutr. 2014 Aug 13;11:38. doi: 10.1186/1550-2783-11-38. eCollection 2014. PMID 25132809
- [Background] Baggett B, Bruckbauer A, Zemel M. Synergistic Effects of Leucine and its Metabolites with Polyphenols on Irisin in Myotubes and Diet-induced Obese Mice. FASEB J. 2013;27:637.11.
- [Background] Huh JY, Dincer F, Mesfum E, Mantzoros CS. Irisin stimulates muscle growth-related genes and regulates adipocyte differentiation and metabolism in humans. Int J Obes (Lond). 2014 Dec;38(12):1538-44. doi: 10.1038/ijo.2014.42. Epub 2014 Mar 11. PMID 24614098
- [Background] Lecker SH, Jagoe RT, Gilbert A, Gomes M, Baracos V, Bailey J, Price SR, Mitch WE, Goldberg AL. Multiple types of skeletal muscle atrophy involve a common program of changes in gene expression. FASEB J. 2004 Jan;18(1):39-51. doi: 10.1096/fj.03-0610com. PMID 14718385
- [Background] Smith HJ, Mukerji P, Tisdale MJ. Attenuation of proteasome-induced proteolysis in skeletal muscle by beta-hydroxy-beta-methylbutyrate in cancer-induced muscle loss. Cancer Res. 2005 Jan 1;65(1):277-83. PMID 15665304
- [Background] Holecek M, Muthny T, Kovarik M, Sispera L. Effect of beta-hydroxy-beta-methylbutyrate (HMB) on protein metabolism in whole body and in selected tissues. Food Chem Toxicol. 2009 Jan;47(1):255-9. doi: 10.1016/j.fct.2008.11.021. Epub 2008 Nov 21. PMID 19056452
- [Background] Kovarik M, Muthny T, Sispera L, Holecek M. Effects of beta-hydroxy-beta-methylbutyrate treatment in different types of skeletal muscle of intact and septic rats. J Physiol Biochem. 2010 Dec;66(4):311-9. doi: 10.1007/s13105-010-0037-3. Epub 2010 Aug 20. PMID 20725872
- [Background] Smith HJ, Wyke SM, Tisdale MJ. Mechanism of the attenuation of proteolysis-inducing factor stimulated protein degradation in muscle by beta-hydroxy-beta-methylbutyrate. Cancer Res. 2004 Dec 1;64(23):8731-5. doi: 10.1158/0008-5472.CAN-04-1760. PMID 15574784
- [Background] Russell ST, Tisdale MJ. Mechanism of attenuation by beta-hydroxy-beta-methylbutyrate of muscle protein degradation induced by lipopolysaccharide. Mol Cell Biochem. 2009 Oct;330(1-2):171-9. doi: 10.1007/s11010-009-0130-5. Epub 2009 Apr 30. PMID 19404720
- [Background] Eley HL, Russell ST, Tisdale MJ. Attenuation of depression of muscle protein synthesis induced by lipopolysaccharide, tumor necrosis factor, and angiotensin II by beta-hydroxy-beta-methylbutyrate. Am J Physiol Endocrinol Metab. 2008 Dec;295(6):E1409-16. doi: 10.1152/ajpendo.90530.2008. Epub 2008 Oct 14. PMID 18854427
- [Background] Hao Y, Jackson JR, Wang Y, Edens N, Pereira SL, Alway SE. beta-Hydroxy-beta-methylbutyrate reduces myonuclear apoptosis during recovery from hind limb suspension-induced muscle fiber atrophy in aged rats. Am J Physiol Regul Integr Comp Physiol. 2011 Sep;301(3):R701-15. doi: 10.1152/ajpregu.00840.2010. Epub 2011 Jun 22. PMID 21697520
- [Background] Supinski GS, Callahan LA. beta-hydroxy-beta-methylbutyrate (HMB) prevents sepsis-induced diaphragm dysfunction in mice. Respir Physiol Neurobiol. 2014 Jun 1;196:63-8. doi: 10.1016/j.resp.2014.02.015. Epub 2014 Mar 12. PMID 24632527
- [Background] Molfino A, Gioia G, Rossi Fanelli F, Muscaritoli M. Beta-hydroxy-beta-methylbutyrate supplementation in health and disease: a systematic review of randomized trials. Amino Acids. 2013 Dec;45(6):1273-92. doi: 10.1007/s00726-013-1592-z. Epub 2013 Sep 22. PMID 24057808
- [Background] Fitschen PJ, Wilson GJ, Wilson JM, Wilund KR. Efficacy of beta-hydroxy-beta-methylbutyrate supplementation in elderly and clinical populations. Nutrition. 2013 Jan;29(1):29-36. doi: 10.1016/j.nut.2012.05.005. Epub 2012 Oct 22. PMID 23085015
- [Background] Gruther W, Benesch T, Zorn C, Paternostro-Sluga T, Quittan M, Fialka-Moser V, Spiss C, Kainberger F, Crevenna R. Muscle wasting in intensive care patients: ultrasound observation of the M. quadriceps femoris muscle layer. J Rehabil Med. 2008 Mar;40(3):185-9. doi: 10.2340/16501977-0139. PMID 18292919
- [Background] Mourtzakis M, Wischmeyer P. Bedside ultrasound measurement of skeletal muscle. Curr Opin Clin Nutr Metab Care. 2014 Sep;17(5):389-95. doi: 10.1097/MCO.0000000000000088. PMID 25023190
- [Background] Tillquist M, Kutsogiannis DJ, Wischmeyer PE, Kummerlen C, Leung R, Stollery D, Karvellas CJ, Preiser JC, Bird N, Kozar R, Heyland DK. Bedside ultrasound is a practical and reliable measurement tool for assessing quadriceps muscle layer thickness. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):886-90. doi: 10.1177/0148607113501327. Epub 2013 Aug 26. PMID 23980134
- [Background] Baldwin CE, Paratz JD, Bersten AD. Diaphragm and peripheral muscle thickness on ultrasound: intra-rater reliability and variability of a methodology using non-standard recumbent positions. Respirology. 2011 Oct;16(7):1136-43. doi: 10.1111/j.1440-1843.2011.02005.x. PMID 21645172
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):642-9. doi: 10.1007/s00134-015-3687-3. Epub 2015 Feb 19. PMID 25693448
- [Background] Grosu HB, Lee YI, Lee J, Eden E, Eikermann M, Rose KM. Diaphragm muscle thinning in patients who are mechanically ventilated. Chest. 2012 Dec;142(6):1455-1460. doi: 10.1378/chest.11-1638. PMID 23364680
- [Background] Ochala J, Gustafson AM, Diez ML, Renaud G, Li M, Aare S, Qaisar R, Banduseela VC, Hedstrom Y, Tang X, Dworkin B, Ford GC, Nair KS, Perera S, Gautel M, Larsson L. Preferential skeletal muscle myosin loss in response to mechanical silencing in a novel rat intensive care unit model: underlying mechanisms. J Physiol. 2011 Apr 15;589(Pt 8):2007-26. doi: 10.1113/jphysiol.2010.202044. Epub 2011 Feb 14. PMID 21320889
- [Background] Biolo G, Fleming RY, Maggi SP, Nguyen TT, Herndon DN, Wolfe RR. Inverse regulation of protein turnover and amino acid transport in skeletal muscle of hypercatabolic patients. J Clin Endocrinol Metab. 2002 Jul;87(7):3378-84. doi: 10.1210/jcem.87.7.8699. PMID 12107253
- [Background] Vesali RF, Cibicek N, Jakobsson T, Klaude M, Wernerman J, Rooyackers O. Protein metabolism in leg muscle following an endotoxin injection in healthy volunteers. Clin Sci (Lond). 2009 Dec 14;118(6):421-7. doi: 10.1042/CS20090332. PMID 19751216
- [Background] Paddon-Jones D, Sheffield-Moore M, Cree MG, Hewlings SJ, Aarsland A, Wolfe RR, Ferrando AA. Atrophy and impaired muscle protein synthesis during prolonged inactivity and stress. J Clin Endocrinol Metab. 2006 Dec;91(12):4836-41. doi: 10.1210/jc.2006-0651. Epub 2006 Sep 19. PMID 16984982
- [Background] Klaude M, Mori M, Tjader I, Gustafsson T, Wernerman J, Rooyackers O. Protein metabolism and gene expression in skeletal muscle of critically ill patients with sepsis. Clin Sci (Lond). 2012 Feb;122(3):133-42. doi: 10.1042/CS20110233. PMID 21880013
- [Background] Essen P, McNurlan MA, Gamrin L, Hunter K, Calder G, Garlick PJ, Wernerman J. Tissue protein synthesis rates in critically ill patients. Crit Care Med. 1998 Jan;26(1):92-100. doi: 10.1097/00003246-199801000-00022. PMID 9428549
- [Background] Latronico N, Fenzi F, Recupero D, Guarneri B, Tomelleri G, Tonin P, De Maria G, Antonini L, Rizzuto N, Candiani A. Critical illness myopathy and neuropathy. Lancet. 1996 Jun 8;347(9015):1579-82. doi: 10.1016/s0140-6736(96)91074-0. PMID 8667865
- [Background] Hsieh LC, Chow CJ, Chang WC, Liu TH, Chang CK. Effect of beta-hydroxy-beta-methylbutyrate on protein metabolism in bed-ridden elderly receiving tube feeding. Asia Pac J Clin Nutr. 2010;19(2):200-8. PMID 20460233
- [Background] Kuhls DA, Rathmacher JA, Musngi MD, Frisch DA, Nielson J, Barber A, MacIntyre AD, Coates JE, Fildes JJ. Beta-hydroxy-beta-methylbutyrate supplementation in critically ill trauma patients. J Trauma. 2007 Jan;62(1):125-31; discussion 131-2. doi: 10.1097/TA.0b013e31802dca93. PMID 17215743
- [Background] Hsieh LC, Chien SL, Huang MS, Tseng HF, Chang CK. Anti-inflammatory and anticatabolic effects of short-term beta-hydroxy-beta-methylbutyrate supplementation on chronic obstructive pulmonary disease patients in intensive care unit. Asia Pac J Clin Nutr. 2006;15(4):544-50. PMID 17077073